CLINICAL TRIAL: NCT03150433
Title: Sleep and Pain in Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Maryland (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00100060; R01HL133327 (NIH)
Record Dates: First submitted 2017-05-03; First posted 2017-05-12 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Sickle Cell Disease; Sleep Disturbance; Pain
MeSH Terms: conditions — Anemia, Sickle Cell; Parasomnias; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be masked to treatment condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral symptom management (Experimental): Five sessions working one-on-one with a study interventionist, either in person or by telephone. Includes monitoring of the individual's sleep pattern, feedback and goals for improving sleep and pain management, and addressing cognitive and emotional strategies for managing sleep and pain.
  Interventions: Behavioral: Behavioral symptom management
- Sickle cell disease management (Other): Five sessions working one-on-one with a study interventionist, either in person or by telephone. Includes monitoring of the individual's sleep pattern, information about sickle cell disease and its management, and information about improving sleep and managing pain.
  Interventions: Other: Sickle cell disease management

INTERVENTIONS:
Behavioral: Behavioral symptom management — Individual sessions focused on behavioral and cognitive strategies for managing sleep disturbance, pain, and other symptoms of sickle cell disease
  Arms: Behavioral symptom management
Other: Sickle cell disease management — Individual sessions focused on understanding and managing sickle cell disease
  Arms: Sickle cell disease management

SUMMARY:
This is a study testing the effects of behavioral sleep interventions on pain and brain function in sickle cell disease.

DETAILED DESCRIPTION:
The investigators propose to examine whether changes in sleep alter pain and pain-related outcomes in adults with Sickle Cell Disease (SCD). As many as 70% of adults with SCD experience various sleep disturbances. Pain and sleep are inter-related, such that pain disturbs sleep and disturbed sleep amplifies pain and increases risk for developing chronic pain. Pain processing occurs in the central nervous system, where nociceptive input can be inhibited or facilitated and which can undergo both functional and structural plasticity. When plasticity results in amplification of pain, this central sensitization (CS) manifests as hyperalgesia, allodynia, and spreading of pain and is an important treatment target in its own right. A growing literature implicates central sensitization in SCD, and the investigators find a strong association between laboratory-evoked CS and sleep disturbance in SCD. The neural substrates involved in pain modulation are often disrupted in chronic pain, likely due to the demands pain places on cognitive resources, and similar effects are seen with chronic insomnia. It remains unclear whether these changes occur in SCD and if improving sleep improves central modulation of pain. The potential for improved sleep to reduce pain and CS requires additional investigation, particularly given the significance of sleep disturbance as a mutable risk factor. The investigators will conduct a randomized trial in which it will be determined whether improvements in sleep reduce pain and alter brain processing of pain and cognitive stimuli. The aims are to determine whether treatment of sleep improves pain outcomes in SCD and to determine whether treatment of sleep alters functional connectivity of cognitive and pain modulatory networks using brain imaging in SCD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sickle cell hemoglobinopathy (Homozygous sickle cell disease, Hemoglobin SC disease, or Sickle/beta-thalassemia);
* Adequate facility with English;
* Stable dosing of medications (if taking) for pain and sleep;
* Reports symptoms of insomnia;
* Reports chronic pain

Exclusion Criteria:

* Cognitive impairment;
* Unstable psychiatric disorder;
* Seizure disorder;
* Positive pregnancy or drug test

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-11-05 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Change in Clinical pain as assessed by the Brief Pain Inventory | baseline and 24 weeks
  Average of 4 items from the Brief Pain Inventory; each rated on a 0 (no pain) to 10 (pain as bad as you can imagine); ratings are made of pain right now, typical pain, worst pain, and least pain during the past week. Total sub-score of 0-40 with higher score indicating more pain.

SECONDARY OUTCOMES:
Change in Clinical pain as assessed by the Brief Pain Inventory | baseline and 36 weeks
  Average of 4 items from the Brief Pain Inventory; each rated on a 0 (no pain) to 10 (pain as bad as you can imagine); ratings are made of pain right now, typical pain, worst pain, and least pain during the past week. Total sub-score of 0-40 with higher score indicating more pain.
Change in Central Sensitization Index | baseline and 12 weeks
  Index of thermal temporal summation, mechanical temporal summation, and aftersensations
Change in functional connectivity/cognitive task | baseline and 12 weeks
  Functional magnetic resonance imaging, functional connectivity during cognitive testing

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Campbell, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers